CLINICAL TRIAL: NCT06613074
Title: Ali Pay Intelligent Navigation Applet-aided Pre-hospital Triage for Non-emergency Medical Service Patients With Acute Ischemic Stroke: A Step-wedge Cluster Randomized Controlled Trial
Brief Title: Ali Pay Intelligent Navigation Applet-aided Pre-hospital Triage for Non-emergency Medical Service Patients With Acute Ischemic Stroke
Acronym: i-Path
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Min Lou, Prof. Dr., Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: i-Path
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-09

CONDITIONS: Acute Ischemic Stroke
Keywords: reperfusion therapy; pre-hospital triage
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ali Pay intelligent navigation applet group (Experimental): Patients in regions with Ali Pay intelligent navigation applet being released would be classified as experimental arm.
  In this arm, patients have access to this applet.
  The intelligent navigation applet comprises of three function modules:
  1. Stroke knowledge public education: information regarding prevention and emergency treatment of stroke would be push to users' mobile phones regularly;
  2. Stroke recognition: questionaires, voice interaction, and facial recognition are employed to identify patients with AIS and large vessel occlusion;
  3. Hospital recommendation: this module combines real-time traffic and average in-hopital delay of each stroke center nearby, recommending the stroke center in which patients are mostly likely to receive reperfusion therapy
- Routine pre-hospital triage (No Intervention): Patients in regions without Ali Pay intelligent navigation applet being released would be classified as control arm.
  In this arm, patients do not have access to this applet.

INTERVENTIONS:
Device: Ali Pay intelligent navigation applet — The intelligent navigation applet comprises of three function modules:
  1. Stroke knowledge public education: information regarding prevention and emergency treatment of stroke would be push to users' mobile phones regularly;
  2. Stroke recognition: questionaires, voice interaction, and facial recognition are employed to identify patients with AIS and large vessel occlusion;
  3. Hospital recommendation: this module combines real-time traffic and average in-hopital delay of each stroke center nearby, recommending the stroke center in which patients are mostly likely to receive reperfusion therapy

SUMMARY:
According to the Bigdata Observatory platform for Stroke of China (BOSC), the proportion of patients with acute ischemic stroke (AIS) receiving intravenous thrombolysis or endovascular treatment in China is 5.64% and 1.45% respectively. One of the important reasons for the low treatment rate is the prolonged pre-hospital and in-hospital delay. Besides, for patients receiving reperfusion therapy, the prolonged pre-treatment delay is associated with unfavorable functional outcomes.

Although tons of efforts have been made to improve the efficiency of emergency medical system in the transportation of patients with AIS, little attention has been paid to patients who arrived at hospitals on their owns, which occupying approximately 2/3 of emergency patients. This leaves a huge gap in the pre-hospital management of patietns with AIS.

Therefore, the investigators plan to develop an intelligent navigation system for patients with AIS. For the convenience of public use, this system was carried on the applet of Ali Pay, which has over 1.1 billion users in China. This system comprises of three functional modules, namely stroke knowledge education, stroke recognition and hospital recommendation. The investigators aim to explore whether this intelligent navigatino system could shorten pre-hospital delay and improve functional outcomes of patients with AIS undergoing reperfusion therapy.

DETAILED DESCRIPTION:
According to the Bigdata Observatory platform for Stroke of China (BOSC), the proportion of patients with acute ischemic stroke (AIS) receiving intravenous thrombolysis or endovascular treatment in China is 5.64% and 1.45% respectively. One of the important reasons for the low treatment rate is the prolonged pre-hospital and in-hospital delay. Besides, for patients receiving reperfusion therapy, the prolonged pre-treatment delay is associated with unfavorable functional outcomes.

Although tons of efforts have been made to improve the efficiency of emergency medical system in the transportation of patients with AIS, little attention has been paid to patients who arrived at hospitals on their owns, which occupying approximately 2/3 of emergency patients. This leaves a huge gap in the pre-hospital management of patietns with AIS.

Therefore, the investigators plan to develop an intelligent navigation system for patients with AIS. For the convenience of public use, this system was carried on the applet of Ali Pay, which has over 1.1 billion users in China. This system comprises of three functional modules, namely stroke knowledge education, stroke recognition and hospital recommendation.The investigators aim to explore whether this intelligent navigatino system could shorten pre-hospital delay and improve functional outcomes of patients with AIS undergoing reperfusion therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as acute ischemic stroke undergoing reperfusion therapy within 24 hours of onset

Exclusion Criteria:

* Patients transported to hospitals via emergency medical service
* Patients with in-hospital stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Modified rankin scale (mRS) scores of 0-2 at 90 days after reperfusion therapy | 90 days

SECONDARY OUTCOMES:
Modified rankin scale (mRS) scores of 0-1 at 90 days after reperfusion therapy | 90 days
Modified rankin scale (mRS) scores of 0-3 at 90 days after reperfusion therapy | 90 days
Ordinal analysis of modified rankin scale (mRS) scores at 90 days after reperfusion therapy | 90 days
Time interval between onset to treatment | 1 day
Time interval between onset to hospital | 1 day
Proportion of patients receiving reperfusion beyond time window | 1 day
  Intravenous thrombolysis: treatment initiated within 4.5 - 9 hours after onset Mechanical thrombectomy: treatment initiated within 6 - 24 hours after onset
Proportion of patients receiving mechanical thrombectomy | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoxing People's Hospital, Shaoxing, Zhejing, China